CLINICAL TRIAL: NCT05766020
Title: Training Listening Skills With the Inclusion of Cognitive Control
Acronym: TRAILS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Astrid Van Wieringen, PhD, Professor, Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S63310
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hearing Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate training group (Experimental): Participants in this group will train immediately for 4 weeks. Afterwards, they will not train for the 8 remaining weeks.
  Interventions: Behavioral: Listen training
- Delayed Training Group (Experimental): Participants in this group will receive delayed training after 4 weeks of no training.
  Interventions: Behavioral: Listen training
- Active control group (Experimental): Participants in this group will perform an active control for 4 weeks, followed by 4 weeks of training.
  Interventions: Behavioral: Listen training

INTERVENTIONS:
Behavioral: Listen training — Auditory skills with the inclusion of cognitive control.

SUMMARY:
Participating in spoken conversation constitutes a multitasking situation with concurrent demands on sensorimotor (auditory, postural) and cognitive functioning (memory, updating, task switching and inhibition). As aging affects multisensory integration and cognitive control, these higher-order processes are likely to put accumulating constraints on listening as adults grow older. By training listening skills (not solely auditory skills), the investigators aim at improving overall communication and quality of life. Moreover, the investigators aim at freeing up cognitive resources in the listen task: the better one gets at a certain domain specific task, the less one needs to draw from other resources and, the more resources are free for another concurrent task. The interdisciplinary approach will inform us about ideal audiological rehabilitation or intervention approaches. Pre-posttests comprise behavioral measures to evaluate listening skills and transfer towards non-trained measures. The training is tablet-based and can be performed at home.

DETAILED DESCRIPTION:
Goals of the study:

* Investigate transfer of listening skills to non-trained listening.
* To develop evidence-based guidelines for clinical audiological rehabilitation.
* Investigate if the inclusion of cognitive control frees up cognitive resources to use for another concurrent task.
* Inform about retention following listening training

All participants will be assessed 4 times, with a 4-week interval in between. Participants in the first arm will perform the training during the first two weeks. 4 weeks after training ended and 8 weeks after training ended, retention of training gains will be assessed. Participants in the second arm will perform the delayed training. This is to control for procedural learning effects. After 4 weeks they will start training for 4 weeks. After training retention of training gains will be assessed after 4 weeks. The third arm will start with active control training (listening to stories) for 4 weeks, followed by training for 4 weeks. After these 8 weeks, retention was measured 4 weeks later. Participants are randomly allocated to a group. The efficacy of training will be determined with a within-subject design (i.e. baseline session outcomes will be compared to the final session outcomes of the randomized control trial.

ELIGIBILITY:
Inclusion Criteria

* Clients who experience listening and communication difficulties.
* Clients must not undergo any audiological rehabilitation (auditory training/hearing aid fitting) during the study.
* Able to operate the training programme as an app on a tablet (e.g. clients have sufficient eyesight to see the exercises; clients must be able to operate the programme).
* At least 18 years old.
* Dutch-speaking, as all training material and counselling questions will be presented in Dutch.

Exclusion Criteria (all groups):

* Severely visually impaired
* Motorically impaired
* Cognitively impaired

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Speech in noise intelligibility | 0 weeks
  LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST) was specifically designed for speech perception in noise assessment in CI users. The test has high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the active training will be an improvement of 2dB on speech perception in noise.
Speech in noise intelligibility | 4 weeks
  LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST) was specifically designed for speech perception in noise assessment in CI users. The test has high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the active training will be an improvement of 2dB on speech perception in noise.
Speech in noise intelligibility | 8 weeks
  LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST) was specifically designed for speech perception in noise assessment in CI users. The test has high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the active training will be an improvement of 2dB on speech perception in noise.
Speech in noise intelligibility | 12 weeks
  LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST) was specifically designed for speech perception in noise assessment in CI users. The test has high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the active training will be an improvement of 2dB on speech perception in noise.
phoneme identification in noise | 0 weeks
  The consonant identification task in noise consisted of 12 Dutch/Flemish vowels presented in an /a/ context. Stimuli were produced by a female speaker. In order not to obtain 100% at the start, stimuli were presented in speech-weighted noise.
phoneme identification in noise | 4 weeks
  The consonant identification task in noise consisted of 12 Dutch/Flemish vowels presented in an /a/ context. Stimuli were produced by a female speaker. In order not to obtain 100% at the start, stimuli were presented in speech-weighted noise.
phoneme identification in noise | 8 weeks
  The consonant identification task in noise consisted of 12 Dutch/Flemish vowels presented in an /a/ context. Stimuli were produced by a female speaker. In order not to obtain 100% at the start, stimuli were presented in speech-weighted noise.
phoneme identification in noise | 12 weeks
  The consonant identification task in noise consisted of 12 Dutch/Flemish vowels presented in an /a/ context. Stimuli were produced by a female speaker. In order not to obtain 100% at the start, stimuli were presented in speech-weighted noise.

SECONDARY OUTCOMES:
The temporal modulation Transfer function | 0 weeks
  With this task, we measure the modulation threshold that listeners need to distinguish between unmodulated and modulated noise, which is related to speech understanding.
The temporal modulation Transfer function | 4 weeks
  With this task, we measure the modulation threshold that listeners need to distinguish between unmodulated and modulated noise, which is related to speech understanding.
The temporal modulation Transfer function | 8 weeks
  With this task, we measure the modulation threshold that listeners need to distinguish between unmodulated and modulated noise, which is related to speech understanding.
The temporal modulation Transfer function | 12 weeks
  With this task, we measure the modulation threshold that listeners need to distinguish between unmodulated and modulated noise, which is related to speech understanding.
Dual-task listening postural control | 0 weeks
  This task aims at identifying the ability to perform two tasks simultaneously. Participants will perform a listening-posture dual-task, where they have to maintain their balance while listening and repeating heard sentences.
Dual-task listening postural control | 4 weeks
  This task aims at identifying the ability to perform two tasks simultaneously. Participants will perform a listening-posture dual-task, where they have to maintain their balance while listening and repeating heard sentences.
Dual-task listening postural control | 8 weeks
  This task aims at identifying the ability to perform two tasks simultaneously. Participants will perform a listening-posture dual-task, where they have to maintain their balance while listening and repeating heard sentences.
Dual-task listening postural control | 12 weeks
  This task aims at identifying the ability to perform two tasks simultaneously. Participants will perform a listening-posture dual-task, where they have to maintain their balance while listening and repeating heard sentences.
Stroop task | 0 weeks
  The Stroop task assesses inhibitory control by requiring participants to identify the color in which a symbol or word is presented while ignoring the word's meaning. Participants were asked to respond to the color of the word while ignoring the written word, which is a color itself.
Stroop task | 4 weeks
  The Stroop task assesses inhibitory control by requiring participants to identify the color in which a symbol or word is presented while ignoring the word's meaning. Participants were asked to respond to the color of the word while ignoring the written word, which is a color itself.
Stroop task | 8 weeks
  The Stroop task assesses inhibitory control by requiring participants to identify the color in which a symbol or word is presented while ignoring the word's meaning. Participants were asked to respond to the color of the word while ignoring the written word, which is a color itself.
Stroop task | 12 weeks
  The Stroop task assesses inhibitory control by requiring participants to identify the color in which a symbol or word is presented while ignoring the word's meaning. Participants were asked to respond to the color of the word while ignoring the written word, which is a color itself.
EAS (Effort Assessment Scale) | 0 weeks
  EAS is a validated scale to measure listening effort. The EAS consists of 6 items that are scored by the client on a 10-point scale, no effort to lots of effort. The EAS questions were translated to Dutch for this study.
EAS (Effort Assessment Scale) | 4 weeks
  EAS is a validated scale to measure listening effort. The EAS consists of 6 items that are scored by the client on a 10-point scale, no effort to lots of effort. The EAS questions were translated to Dutch for this study.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | 0 weeks
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | 4 weeks
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid van Wieringen, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Experimental ORL, Dept Neurosciences, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Background] van Wieringen A, Wouters J. Natural vowel and consonant recognition by Laura cochlear implantees. Ear Hear. 1999 Apr;20(2):89-103. doi: 10.1097/00003446-199904000-00001. PMID 10229511
- [Background] van Wieringen A, Wouters J. LIST and LINT: sentences and numbers for quantifying speech understanding in severely impaired listeners for Flanders and the Netherlands. Int J Audiol. 2008 Jun;47(6):348-55. doi: 10.1080/14992020801895144. PMID 18569107
- [Background] Noble W. Hearing, hearing impairment, and the audible world: a theoretical essay. Audiology. 1983;22(4):325-38. doi: 10.3109/00206098309072793. PMID 6615338
- [Background] Alhanbali S, Dawes P, Lloyd S, Munro KJ. Self-Reported Listening-Related Effort and Fatigue in Hearing-Impaired Adults. Ear Hear. 2017 Jan/Feb;38(1):e39-e48. doi: 10.1097/AUD.0000000000000361. PMID 27541332
- [Derived] Van Wilderode M, Van Humbeeck N, Krampe RT, van Wieringen A. Enhancing Speech Perception in Noise Through Home-Based Competing Talker Training. Ear Hear. 2025 Jul-Aug 01;46(4):856-870. doi: 10.1097/AUD.0000000000001631. Epub 2025 Feb 10. PMID 39924678